CLINICAL TRIAL: NCT07173283
Title: Evaluation of the Impact of a Peer Mentorship Program on the Professional Integration of Newly Graduated Occupational Therapists: The MenTOras Program
Brief Title: Peer Mentorship Program for Newly Graduated Occupational Therapists in Aragón (MenTOras)
Acronym: MenTOras
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sandra León-Herrera, PhD Student, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SL_CEIN_2025_16
Record Dates: First submitted 2025-08-29; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Professional Integration of Newly Graduated Occupational Therapists; Peer Mentorship in Health Professions; Early Career Transition and Professional Identity
Keywords: Occupational Therapy; Peer Mentorship; Professional Development; Newly Graduated Health Professionals; Early Career Support; Professional Identity; Job Satisfaction; Spain; Pilot Study
MeSH Terms: interventions — Occupational Therapists

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental, prospective pilot study in which all participants receive the MenTOras peer mentorship program. There is no control group, and outcomes are assessed at baseline, after the intervention, and at six-month follow-up.
Masking Description: Neither participants, nor researchers, nor evaluators are blinded; this is an educational and mentoring program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Mentorship Program for Early-Career Occupational Therapists (Other): This arm involves participation in the MenTOras peer mentorship program, a structured three-month intervention designed for newly graduated occupational therapists in Aragón, Spain. Each participant is paired with an experienced occupational therapist who provides professional guidance, reflective practice, and emotional support. Mentor-mentee pairs engage in at least six structured sessions (online or in person), complemented by COPTOA-organized training workshops. The program is organized in three phases-initiation (goal-setting and rapport building), development (professional identity, problem-solving, and emotional support), and closure (reflection and planning for continued growth). Outcomes focus on professional integration, self-confidence, and mentees' well-being, as well as mentors' reciprocal learning.
  Interventions: Other: MenTOras: Peer Mentorship Program for Newly Graduated Occupational Therapists

INTERVENTIONS:
Other: MenTOras: Peer Mentorship Program for Newly Graduated Occupational Therapists — The MenTOras intervention is a structured peer mentorship program designed for newly graduated occupational therapists in Aragón, Spain. The program pairs early-career occupational therapists (mentees, graduated within the past two years) with experienced colleagues (mentors, with at least five years of practice). Over approximately three months, each mentor-mentee pair participates in at least six structured sessions (online or in person). Sessions follow three phases-initiation, development, and closure-focusing on professional identity, reflective practice, emotional support, and skill integration. Mentors receive orientation and guidance to ensure program consistency. COPTOA also offers topic-specific training to address emerging professional needs. The intervention aims to foster professional integration, enhance self-confidence, and promote well-being among new occupational therapists, while strengthening professional cohesion and retention.
  Other Names: Peer Mentoring for Occupational Therapists in Aragón

SUMMARY:
This study evaluates the MenTOras program, a structured peer mentorship intervention designed for newly graduated occupational therapists in Aragón, Spain. The transition from university to professional practice can be challenging, and many new occupational therapists face isolation, limited guidance, and uncertainty about their professional role.

The MenTOras program connects newly graduated occupational therapists (mentees) with more experienced colleagues (mentors). Over a three-month period, mentor-mentee pairs participate in at least six structured sessions, either online or in person. These sessions are designed to support professional integration, strengthen self-confidence, promote reflective practice, and provide emotional support.

The study uses a mixed-methods approach. Quantitative data are collected before the program, after completion, and six months later to assess perceived professional integration, emotional well-being, and professional confidence. In addition, qualitative interviews with a subset of participants explore their experiences in greater depth.

By fostering peer support, MenTOras aims to improve the early career experience of occupational therapists and provide a model for sustainable mentoring practices within the profession.

DETAILED DESCRIPTION:
The MenTOras project is a pilot study developed in response to the lack of structured mentorship opportunities for occupational therapists in Spain. International research highlights that mentorship improves professional integration, emotional well-being, and retention within health professions, but formal mentorship programs for occupational therapists in Spain are scarce.

Study Design This is a prospective, mixed-methods, quasi-experimental pilot study without a control group, using a successive cohort design. Approximately 20 mentor-mentee pairs (40 participants in total) will be recruited. Occupational therapists who have graduated within the past two years will be eligible as mentees, while mentors must have at least five years of professional experience. All participants must be members of the Colegio Profesional de Terapeutas Ocupacionales de Aragón (COPTOA).

Intervention

The MenTOras program lasts about three months and consists of three phases:

* Initiation: establishing rapport, setting expectations, and defining goals.
* Development: structured mentoring sessions focusing on professional identity, reflective practice, and emotional support.
* Closure: reflection on progress and planning next steps.

Pairs will participate in at least six mentoring sessions, adapted to the mentee's needs and professional area. Mentors receive orientation and ongoing support from the research team. COPTOA will also organize additional training sessions on relevant professional topics.

Outcomes and Data Collection Data will be collected at three time points: baseline (pre-program), post-program, and six-month follow-up. Quantitative measures include the mentees' perceived professional integration, emotional well-being, and professional self-confidence, as well as satisfaction with the program. Mentors will report their perceptions of mentee growth, satisfaction with the mentoring process, and their own learning.

Additionally, semi-structured interviews will be conducted with a subset of participants to explore the mentoring experience, perceived benefits, and suggestions for improvement.

Analysis Quantitative data will be analyzed using descriptive and inferential statistics, including repeated measures analyses. Qualitative data will be analyzed thematically using established frameworks to capture participants' experiences and recommendations. The integration of both data types will provide a comprehensive understanding of the program's feasibility, acceptability, and impact.

Significance This pilot study seeks to provide evidence on the feasibility and effectiveness of a peer mentorship program for newly graduated occupational therapists in Spain. If successful, MenTOras could be expanded to other regions and serve as a model for structured mentoring programs across health professions. The findings may also inform policies aimed at improving workforce retention, professional identity, and the integration of occupational therapists into healthcare and social systems.

ELIGIBILITY:
Inclusion Criteria (Mentees - Recently graduated occupational therapists):

* Completed a degree in Occupational Therapy within the past 2 years.
* May or may not be currently employed in the profession.
* Registered member of the Aragon Professional Association of Occupational Therapists (COPTOA).

Inclusion Criteria (Mentors - Experienced occupational therapists):

* Minimum of 5 years of clinical or community-based practice in occupational therapy.
* Actively practicing at the time of enrollment.
* Registered member of COPTOA.

Exclusion Criteria (applies to both groups unless otherwise specified):

* For mentors: occupational therapists who are no longer actively practicing.
* For all participants: current involvement in another mentorship program or structured training initiative with overlapping objectives.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in perceived professional integration of newly graduated occupational therapists | Baseline (pre-program), immediately post-intervention (3 months), and 6-month follow-up.
  Definition: Newly graduated occupational therapists' perceived integration into the profession was assessed using study-specific items.
  Instrument:
  5-point Likert scale items (1 = strongly disagree, 5 = strongly agree)
  Areas assessed: professional confidence, sense of belonging to the occupational therapy community, perceived usefulness of the mentoring experience
  Interpretation:
  Higher scores indicate greater perceived professional integration, including stronger role confidence, a stronger sense of belonging, and a more positive perception of the mentoring process.
  Example questionnaire items:
  "I feel confident in my role as an occupational therapist." "I feel actively part of the occupational therapy professional community." "I feel that I have someone to rely on for my professional development."

SECONDARY OUTCOMES:
Change in emotional well-being | Baseline, immediately post-intervention, and 6-month follow-up.
  Definition: Participants' emotional well-being was assessed before and after the mentoring program.
  Instrument:
  Study-specific Likert items rated on a 5-point scale (1 = strongly disagree, 5 = strongly agree)
  Includes perceived emotional stability, coping with professional challenges, and overall satisfaction with mentoring
  Interpretation:
  Higher scores indicate better emotional well-being, greater stability, and higher confidence in facing professional challenges.
  Example questionnaire items:
  "I feel emotionally prepared to face the challenges of my professional practice." "The mentoring helped me adapt better to the work environment." "How would you rate the impact of the program on your emotional well-being?" (Likert 1-5)
Change in professional self-confidence | Baseline, immediately post-intervention, and 6-month follow-up.
  Definition: Participants' confidence in their professional skills and decision-making was measured using study-specific items.
  Instrument:
  Likert-type items (1 = strongly disagree, 5 = strongly agree)
  Includes categorical items on self-reported improvement in professional confidence
  Interpretation:
  Higher scores indicate greater confidence in clinical decision-making and professional competence.
  Example questionnaire items:
  "I trust my ability to make appropriate clinical decisions." "Has your professional self-confidence improved after participating in the program?" (Categories: greatly improved, somewhat improved, unchanged, worsened)
Participant satisfaction with the mentorship program | Immediately post-intervention.
  Definition: Assessment of participants' perceived usefulness and satisfaction with the mentoring experience.
  Instrument:
  Likert-type items (1-5) measuring:
  * Quality of the mentor-mentee relationship
  * Usefulness of mentoring sessions
  * Overall satisfaction with the program
  * Open-ended questions on benefits and suggested improvements
  Interpretation:
  Higher scores reflect greater satisfaction, perceived program benefit, and willingness to participate again or recommend the program.
  Example questionnaire items:
  "The relationship with my mentee/mentor was positive." "I would like to repeat the experience." "Which aspects of the program have been most beneficial for you as a mentor?" (open-ended)

OTHER OUTCOMES:
Mentor-reported outcomes | Immediately post-intervention and at 6-month follow-up.
  Instrument: Mentor Impact Questionnaire 5-point Likert scale (1 = strongly disagree, 5 = strongly agree) on:
  * Mentee professional growth (emotional well-being, usefulness of mentorship)
  * Mentor professional development (clinical confidence, emotional readiness, engagement in the occupational therapy community)
  * Program satisfaction (quality of relationship, willingness to participate again)
  Categorical items: Yes/No/Moderate Open-ended questions on challenges, benefits, and suggestions for improvement
  Interpretation:
  Higher scores indicate greater perceived positive impact on mentees, mentor professional development, and overall satisfaction with the program.
Qualitative insights from semi-structured interviews | 4-6 weeks after program completion.
  Objective: Explore experiences and perceptions of both mentors and mentees, including:
  * Professional identity development
  * Emotional support
  * Challenges and recommendations for program improvement
  Method:
  Thematic analysis of open-ended questionnaire responses and interviews to complement quantitative data

CONTACTS AND LOCATIONS:
Overall Officials: Sandra León-Herrera, PhD student, Principal Investigator — Universidad de Zaragoza; Marta Marín-Berges, Adjunct Professor, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Colegio Profesional de Terapeutas Ocupacionales de Aragón (COPTOA), Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. Findings will be reported only in aggregated, anonymized form in peer-reviewed scientific publications and conference presentations.